CLINICAL TRIAL: NCT02123212
Title: Birth-Cohort Evaluation to Advance Screening and Testing for Hepatitis C
Acronym: Best-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Opinion Research Center (Other)
Collaborators: NORC at the University of Chicago (Other); University of Alabama at Birmingham (Other); Henry Ford Health System (Other); Icahn School of Medicine at Mount Sinai (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. David Rein, Principal Research Scientist, National Opinion Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 527-11 SC; 6960 (Other: NORC)
Record Dates: First submitted 2014-04-22; First posted 2014-04-25 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C; Chronic Hepatitis C
Keywords: Hepatitis C; Chronic Hepatitis C; Screening
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mt. Sinai (Experimental): Cluster randomization with EHR Alert intervention
  Interventions: Other: EHR Alert
- Henry Ford Health System (Experimental): Simple randomization with mailer intervention
  Interventions: Other: Mailer
- University of Alabama, Birmingham (Experimental): Crossover randomization with in-person recruitment intervention
  Interventions: Other: In-person recruitment

INTERVENTIONS:
Other: Mailer — Henry Ford intentifies patients meeting birth cohort screening criteria and then sends mailers to those individuals. Mailers contained HCV guidelines, the importance of screening, laboratory slips and locations for patients to act directly on their own behalf. If patients do not respond to the initial mailer, Henry Ford sends additional mailers.
  Arms: Henry Ford Health System
Other: In-person recruitment — UAB used study coordinators to actively screen and recruit patients who met the inclusion criteria for birth-cohort screening. Study coordinators were located at two internal medicine clinics, where they approached eligible participants in person. A control group was pulled from an additional two internal medicine clinics, which screened using a risk-based strategy. A cross-over approach was used, so that the intervention and control clinics switched at the midpoint of data collection, allowing all four clinics to participate in both arms of the study.
  Arms: University of Alabama, Birmingham
Other: EHR Alert — EHR include a Best Practice Alert (BPA) prompting the Medical Assistant and/or clinican to order a Hepatitis C lab test for patients in the birth cohort.
  Arms: Mt. Sinai

SUMMARY:
The Birth-Cohort Evaluation to Advance Screening and Testing for Hepatitis C (BEST-C) compares the effectiveness of the birth cohort HCV screening strategy with the current risk-based screening approach to detect previous unidentified persons with viral hepatitis C who receive health care in primary systems.

The study involved three clinical sites, The University of Alabama, Birmingham; The Henry Ford Health System; and the Mount Sinai Medical Center, each of which developed an independent intervention to experimentally compare the number of positive Hepatitis C Virus (HCV) diagnoses found using the birth-cohort screening approach with that found using traditional risk-based screening, or standard of care strategies. Birth cohort testing is defined as the systematic recommendation of HCV antibody testing to any persons born during the years of 1945 to 1965 who do not have clinically documented evidence of a prior antibody test without regards to the patient's stated risk of exposure to the virus.

DETAILED DESCRIPTION:
The Birth-Cohort Evaluation to Advance Screening and Testing for Hepatitis C (BEST-C) compares the effectiveness of the birth cohort HCV screening strategy with the current risk-based HCV screening approach to detect previously unidentified persons with viral hepatitis C who receive health care in primary care systems.

BEST-C funded sites to implement birth-cohort testing in a clinic sample of primary care patients using an experimental design to compare the effect of birth-cohort testing on testing rates and identified prevalence between a case and a control sample. Additional data will be collected to assess linkage to care for those testing positive, feasibility, and acceptance of the new strategy by medical staff, cost effectiveness, and patient impact. The sites used three models to measure the net effect of change:

One site used study coordinators to actively screen and recruit patients who met the inclusion criteria for birth-cohort screening. Study coordinators were located at two internal medicine clinics, where they approached eligible participants in person. A control group was pulled from an additional two internal medicine clinics, which screened using a risk-based strategy. A cluster randomized cross-over approach was used, so that the intervention and control clinics switched at the midpoint of data collection, allowing all four clinics to participate in both arms of the study.

A second site reached out directly to the patient using direct communication through the mail. Mailers contained HCV guidelines, the importance of screening, laboratory slips and locations for patients to act directly on their own behalf. This site used simple randomization of patients who used the health system in the past, met the definition of birth-cohort membership (born during 1945 to 1965) and had not previously tested positive for hepatitis C. The patients received up to 5 mailings including prepaid, lab registration forms that they were instructed to bring to an affiliated lab location for testing.

A third site implemented a physican best practice alert into the Epic electronic health record system of their clinic setting. This site had the pop-ups enabled for Medical Assistants (MAs) who were asked to pend the lab to the order in the chart for the clinician. When MAs open the chart of an arrived, untested patient, they are alerted to pend the Hepatitis C antibody test order when entering patient vitals prior to the patient seeing the physician. When the clinician subsequently opened the same patient chart, the lab order was present in the orders section of the chart for signature and execution or deletion depending on the circumstances of the patient encounter. As a back-up pathway alerted the physician directly in the event that the MA bypassed or did not open the prompt. This alert details the CDC recommendations for age-based screening and links to the proper Hepatitis C antibody test order and diagnosis code for them to address with the patient.

This site used a cluster randomized experimental design in which physicians and MA's from specific primary care practices were consented into the study. Experimental clusters received an education about HCV testing and the implemented best practice alert. Control clusters received only education about HCV testing.

ELIGIBILITY:
Inclusion Criteria:

* Born 1945-1965

Exclusion Criteria:

* Prior diagnosis of Hepatitis C

Ages: 47 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29607 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Positive Hepatitis C Test | Up to 16 weeks
  Positive diagnosis on a Hepatitis C test

SECONDARY OUTCOMES:
Tested for Hepatitis C | Up to 16 weeks
  Patient received a test for Hepatitis C

CONTACTS AND LOCATIONS:
Overall Officials: David B Rein, Ph.D., Principal Investigator — NORC at the University of Chicago
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Henry Ford Health System, Detroit, Michigan
  - Mt. Sinai Medical Center, New York, New York

REFERENCES:
- [Background] Rein DB, Smith BD, Wittenborn JS, Lesesne SB, Wagner LD, Roblin DW, Patel N, Ward JW, Weinbaum CM. The cost-effectiveness of birth-cohort screening for hepatitis C antibody in U.S. primary care settings. Ann Intern Med. 2012 Feb 21;156(4):263-70. doi: 10.7326/0003-4819-156-4-201202210-00378. Epub 2011 Nov 4. PMID 22056542
- [Background] Smith BD, Yartel AK, Krauskopf K, Massoud OI, Brown KA, Fallon MB, Rein DB. Hepatitis C virus antibody positivity and predictors among previously undiagnosed adult primary care outpatients: cross-sectional analysis of a multisite retrospective cohort study. Clin Infect Dis. 2015 Apr 15;60(8):1145-52. doi: 10.1093/cid/civ002. Epub 2015 Jan 16. PMID 25595745
- [Background] Jewett A, Garg A, Meyer K, Wagner LD, Krauskopf K, Brown KA, Pan JJ, Massoud O, Smith BD, Rein DB. Hepatitis C virus testing perspectives among primary care physicians in four large primary care settings. Health Promot Pract. 2015 Mar;16(2):256-63. doi: 10.1177/1524839914532291. Epub 2014 Apr 28. PMID 24776636
- [Derived] Federman AD, Kil N, Kannry J, Andreopolous E, Toribio W, Lyons J, Singer M, Yartel A, Smith BD, Rein DB, Krauskopf K. An Electronic Health Record-based Intervention to Promote Hepatitis C Virus Testing Among Adults Born Between 1945 and 1965: A Cluster-randomized Trial. Med Care. 2017 Jun;55(6):590-597. doi: 10.1097/MLR.0000000000000715. PMID 28288075